CLINICAL TRIAL: NCT00189306
Title: An Open-label Study to Evaluate the Safety and Long-Term Clinical Efficacy of Imiquimod 5% Cream Applied Once Daily 7 Days Per Week for 6 Weeks in the Treatment of Superficial Basal Cell Carcinoma
Brief Title: Open-label Study to Evaluate Clearance of Superficial Basal Cell Carcinoma After Use of Imiquimod 5% Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Medical Director, Graceway Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1413-IMIQ
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2008-11-26 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: Superficial Basal Cell Carcinoma; Aldara
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aldara (Experimental): Aldara (imiquimod) cream 5% applied 7 times per week for 6 weeks
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Aldara (imiquimod) 5% cream - 250 mg / packet - once daily 7 days per week for 6 weeks
  Other Names: Aldara (imiquimod) 5% cream - 250 mg / packet

SUMMARY:
An open-label study to evaluate the safety and the ability of Imiquimod 5% cream, applied topically, to clear superficial basal cell carcinoma and to keep it clear for 5 years of follow-up.

DETAILED DESCRIPTION:
Evaluate the long-term sustained clearance rate, defined as the proportion of those subjects clinically clear of basal cell carcinoma (BCC) at the treated superficial BCC (sBCC) target tumor site at the 12-week posttreatment visit who remain clear during a 5 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 previously untreated superficial basal cell carcinoma tumor
* Minimum tumor size 0.5 cm2 and maximum diameter of 2.0 cm

Exclusion Criteria:

* Evidence of clinically significant, unstable medical conditions
* Cannot have recent use of topical steroids or retinoids in the treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2001-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Lee, Dr., Study Director — Graceway Pharmaceuticals
Locations (18):
- Australia (13):
  - Medical Centre, Concord Hospital, Concord, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Skin Centre, Benowa, Queensland
  - South East Dermatology Centre, Carina Heights, Queensland
  - 105 Fulham Road, Gulliver, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Center, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Western Hospital, Footscray, Victoria
  - Austin & Repartriation Hospital, Heidelburg, Victoria
  - Freemantle Dermatology, Fremantle, Western Australia
  - 158 South Terrace, Perth, Western Australia
  - Subiaco Clinic, Subiaco, Western Australia
- New Zealand (5):
  - 103A Mountain Road, Epsom, Auckland
  - Birthcare Building, Parnell, Auckland
  - Colombo Mansions, Christchurch
  - Dermatology Practice, Christchurch
  - Skin Institute Limited, Takapuna

REFERENCES:
- [Result] Quirk C, Gebauer K, Owens M, Stampone P. Two-year interim results from a 5-year study evaluating clinical recurrence of superficial basal cell carcinoma after treatment with imiquimod 5% cream daily for 6 weeks. Australas J Dermatol. 2006 Nov;47(4):258-65. doi: 10.1111/j.1440-0960.2006.00313.x. PMID 17034468
- [Result] Quirk C, Gebauer K, De'Ambrosis B, Slade HB, Meng TC. Sustained clearance of superficial basal cell carcinomas treated with imiquimod cream 5%: results of a prospective 5-year study. Cutis. 2010 Jun;85(6):318-24. PMID 20666194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in 18 study centers: 13 in Australia and 5 in New Zealand. The first subject entered this study on 27 March 2001; the last clinic visit was on 20 April 2007 and the last subject status determination (subject lost to follow-up) was on 27 April 2007.
Pre-assignment Details: There were 169 subjects enrolled at 18 study centers in Australia and New Zealand.
Groups:
- Aldara: Aldara (imiquimod) cream 5%
Period: Treatment Period
Arm/Group | Aldara
Started | 169
Completed | 164 (5 subjects discontinued during treatment - 4 subjects returned for the Posttreatment Period)
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Period: Posttreatment Period
Arm/Group | Aldara
Started | 169 (5 of the 169 discontinued, but 4 returned for the Posttreatment Period)
Completed | 157 (11 subjects discontinued during the 12-week Posttreatment Period)
Not Completed | 12
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Noncompliance | 1
Not completed — Target lesion excised | 1
Not completed — Protocol Violation | 1
Not completed — Evidence of Superficial Basal Cell Ca | 5
Not completed — Local skin reaction/sign | 1
Period: Long-Term Follow-up
Arm/Group | Aldara
Started | 157
Completed | 119
Not Completed | 38
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Intercurrent disease | 2
Not completed — Lost to Follow-up | 9
Not completed — Evidence of Superficial Basal Cell Ca | 20

BASELINE CHARACTERISTICS:
Arm/Group | Aldara
Number analyzed (Participants) | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 130
  >=65 years | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 96
Region of Enrollment [Number; unit: participants]
  Australia | 123
  New Zealand | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Clearance Rate of Superficial Basal Cell Carcinoma (sBCC)
Description: Number of participants clinically clear of superficial basal cell carcinoma at the treated target tumor site at the 12-week posttreatment visit (ie, initial clearance rate) who remain clear during a 5 year follow-up period.
Time Frame: 5 years
Population: 2 data sets: ITT - all enrolled subjects and PP - ITT subjects free from major protocol violations and applied at least 60% of doses required
Measure: Number; unit: participants
Arm/Group | Aldara
Number analyzed (Participants) | 157
participants | 119

2. Secondary Outcome: Number of Participants Cleared of Superficial Basal Cell Carcinoma at 12 Weeks
Description: Number of participants cleared at 12 weeks(the number of subjects with no clinical evidence of superficial basal cell carcinoma at the target tumor site at the 12-week posttreatment visit)
Time Frame: 12 week posttreatment visit
Population: Two data sets were analyzed: intent-to-treat (ITT), consisting of all enrolled subjects and per-protocol (PP), consisting of ITT subjects who were free from major protocol violations, and who applied at least 60% of the doses required by the dosing regimen.
Measure: Number; unit: participants
Arm/Group | Aldara
Number analyzed (Participants) | 169
participants | 159

ADVERSE EVENTS:
Time Frame: Adverse events were reported from post prestudy visit to throughout the treatment and posttreatment period (up to week 12). Serious Adverse Events were recorded throughout the follow-up period (up to the 60 month visit).
Arm/Group | Aldara
Serious Adverse Events (participants affected / at risk) | 23/169
Other Adverse Events (participants affected / at risk) | 130/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aldara (N=169)
Embolism pulmonary (Vascular disorders) | 1 (1)
Non-hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Excision BCC R forehead (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bleeding post colonoscopy (Surgical and medical procedures) | 1 (1)
Transient ischaemic attack (Vascular disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4)
Cholecyctitis (Hepatobiliary disorders) | 1 (1)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (General disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (4)
Goitre (Endocrine disorders) | 1 (1)
Bladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chronic renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aldara (N=169)
Application site reaction (Skin and subcutaneous tissue disorders) | 100 (100)
Headache (Nervous system disorders) | 23 (23)
Pain (General disorders) | 9 (9)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No